CLINICAL TRIAL: NCT05888298
Title: Proximal and Distal Approach GON RFT in Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, director, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GONRFT
Record Dates: First submitted 2023-02-10; First posted 2023-06-05 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Migraine Disorders; Headache Migraine Chronic
Keywords: greater occipital nerve block; radiofrequency
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal block (Active Comparator): GON block is performed at C2 vertebra level
  Interventions: Procedure: Greater occipital nerve radiofrequency
- Distal block (Other): GON block is performed at occipital protuberence
  Interventions: Procedure: Greater occipital nerve radiofrequency

INTERVENTIONS:
Procedure: Greater occipital nerve radiofrequency — Greater nerve block and radiofrequency will be performed at the C2 vertebra level or occipital protuberance

SUMMARY:
Greater occipital nerve pulsed radiofrequency therapy is used in the treatment of migraine. This method is applied at the level of the proximal c2 vertebra and by approaching the nerve from the distal 1/3 medial of the occipital protuberant. The investigators aimed to compare the effectiveness of these two methods.

DETAILED DESCRIPTION:
Greater occipital nerve (GON) pulsed radiofrequency application is used in migraine headaches. The procedure is applied by approaching the occipital nerve trace with a radiofrequency needle, giving a pulsed radiofrequency current for 4 minutes, and then injecting 2.5 cc bupivacaine and saline. There are two types of applications. In the proximal/central approach, the injection is administered to the occipital nerve between the semispinalis capitis muscle and the obliquus capitis inferior, under ultrasound guidance, while in the distal approach, it is administered 1/3 cm medial to the occipital protuberant with a blind technique.

The investigators aim to compare the treatment response at 1 and 3 months between two patient groups treated with both methods. For this purpose, The investigators planned to follow up with 60 patients. GON RF will be performed with a proximal approach to half of the patients and a distal approach to the other half. Pain levels will be measured on the Visual Analogue Scale (VAS) in the 1st and 3rd months after the procedure. Migraine Disability Index (MIDAS) will be applied to the patients in the 1st week and 3rd month after the procedure. Thus, it will be determined whether there is a difference between the approaches in terms of pain palliation.

Patients who have undergone the procedure will be found from their file records and called by phone, when they come to the control, face to face and 1-3. In the months, the scales will be filled by calling by phone.

ELIGIBILITY:
Inclusion Criteria:

* Primary migraine hedache, first interventional treatment for headache

Exclusion Criteria:

* Preganancy, malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-22 (Estimated); Study Completion 2023-12-28 (Estimated)

PRIMARY OUTCOMES:
The MIDAS (Migraine Disability Assessment) questionnaire | Change from Baseline MIDAS at 3 months
  The MIDAS (Migraine Disability Assessment) questionnaire was put together to help you measure the impact the headaches. The information on this questionnaire is also helpful the primary care provider to determine the level of pain and disability caused by your headaches.
VAS Visual analog scale | Change from Baseline MIDAS at 3 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Yuruk, Study Director — Diskapi TRH
Locations (2):
- Turkey (Türkiye) (2):
  - Diskapi Training and Research Hospital, Ankara
  - Dişkapi Reserch and Education Hospital, Ankara